CLINICAL TRIAL: NCT01341106
Title: Induction of Fibrosis Regression on Patients With Chronic Hepatitis B Infection
Acronym: INFIRE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: insufficient patient numbers have been recruited
Sponsor: RWTH Aachen University (Other)
Collaborators: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CTC-A 11-018; 2010-019884-12 (EudraCT Number); 11-018 (Other: CTC-A)
Record Dates: First submitted 2011-04-20; First posted 2011-04-25 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis B, Chronic; Liver Fibrosis
Keywords: chronic hepatitis B; liver fibrosis; treatment with Entecavir
MeSH Terms: conditions — Hepatitis B, Chronic; Liver Cirrhosis | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm (Experimental): Patients will be treated with entecavir
  Interventions: Drug: Treatment with entecavir(Baraclude®)

INTERVENTIONS:
Drug: Treatment with entecavir(Baraclude®) — Patient will be daily treated with 1 tablet of entecavir per oral

SUMMARY:
This study will examine whether 12 month treatment with entecavir(Baraclude®) has an effect on changes of liver stiffness measurement (LSM) and of hyaluronan measurement in patients with chronic hepatitis B infection.

DETAILED DESCRIPTION:
Patients with chronic hepatitis B infection and relevant liver fibrosis will be treated with entecavir during 5 years or until anti-HBs seroconversion or 6-12 months after anti-HBe seroconversion and HBeAg loss. There are 9 visits during treatment for each patient. At all visits, each patient will consent to give 20 ml blood sample for study examination and 40 ml blood sample for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* chronic hepatitis B infection with detectable HBV (hepatitis B virus)-DNA at baseline
* results of a current liver biopsy (date of liver biopsy must not be longer than 3 months as date of screening visit)
* detection of relevant liver fibrosis in liver histology after percutaneous or laparoscopic biopsy (histologically ≥ F2) after estimation by an experienced pathologist in the liver pathology and sufficient evaluability of the biopsy (usually evaluation of portal at least 8 fields)
* Therapy indication according to current guidelines cHBV infection ( any virus replication in the presence of liver cirrhosis, or detection of HBV-DNA ≥ 2000 IU / ml and/or liver histology with inflammatory Grade ≥2 / fibrosis stage 2 and presence of ALT <5 x ULN)
* non-pregnant and non-breastfeeding women, who fitful one of following criteria: * post-menopausal (12 months natural amenorrhea or 6 months amenorrhea with serum FSH (follicle stimulating hormone)> 40mlU/ml)

  * 6 weeks after surgical sterilization by bilateral tubal transection or after bilateral oophorectomy with or without hysterectomy
  * Correct application of two methods of sure contraception (any combination of a hormonal contraceptive (the pill, hormone IUD (intrauterine device), Depo-Provera, Implanon, contraceptive patch or vaginal ring) or IUD with a barrier contraceptive with spermicide (diaphragm, cervical cap, LEA contraceptive, female condoms or condom)or a spermicide.
  * Sexual abstinence for 2 weeks before the first administration of the study medication, during the study period and after the study during 30 days (time of elimination of study medication)
  * Patients, who have only female sexual partners
  * Male partner of a female patient, who before study inclusion, sterile and only one sexual partner of this female patient is
* Patients willing and able to complete the requirements of this study

Exclusion Criteria:

* anamnestic known hypersensitivity to Baraclude® or its ingredients or to drugs with similar chemical structure
* Participation of patients in another clinical study within last 4 weeks prior to the inclusion or simultaneous participation in another clinical study
* anamnestic known substance dependance or another diseases, which not allowed persons to understand essence and importance and possible consequences of the trial
* lack of cooperation and informed consent
* co-infection with hepatitis C, hepatitis D or HIV
* detection of hepatocellular carcinoma
* serious, chronic disease with an estimated prognosis for survival shorter than the study period of 5 years
* every previous therapy with lamivudine or telbivudine or previous therapy with other antiviral substance within last 6 months before study inclusion
* contraindications to the use of entecavir
* creatinine clearance <50 ml / min and / or need for hemodialysis
* MELD score >15 points and / or detection of ascites

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-04; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Changes of liver stiffness measurement (LSM) and hyaluronan measurement in blood | 12 Month
  Changes of liver stiffness measurement (LSM) and hyaluronan measurement in blood will be checked as markers of fibrous tissue in the liver after treatment with entecavir(Baraclude®) within 12 month.

SECONDARY OUTCOMES:
Changes on Pro-Collagen-III-N-Peptid, Tissue Inhibitor of Metalloproteinases (TIMP-1) and Chitinase-3-like protein 1(YKL-40) in serum | 12 Month
  Changes on Pro-Collagen-III-N-Peptid, Tissue Inhibitor of Metalloproteinases (TIMP-1) and Chitinase-3-like protein 1(YKL-40) in serum will be checked after 12 month treatment.
Sensitivity and specificity of non-invasive marker at the baseline in comparison to liver biopsy as a gold standard | 12 Month
  Non-invasive marker(liver stiffness measurement(LSM) with FibroScan and serum parameter(hyaluronan measurement, Pro-Collagen-III-N-Peptid, Tissue Inhibitor of Metalloproteinases(TIMP-1) and Chitinase-3-like protein 1(YKL-40))) at the baseline will be compared with results of liver biopsy as gold standard after treatment with entecavir(Baraclude®) within 12 month.
Changes on FibroScan-measurement (LSM) and serum parameter | 6,12,18,24,36,48 and 60 month
  Changes on FibroScan-measurement (LSM) and serum parameter (hyaluronan measurement, Pro-Collagen-III-N-Peptid, Tissue Inhibitor of Metalloproteinases(TIMP-1) and Chitinase-3-like protein 1(YKL-40))) will be checked at timepoints of 6,12,18,24,36,48 and 60 month after treatment with entecavir(Baraclude®) within 12 month.
Decrease of hepatitis B virus-DNA and quota of patients with non-detectable hepatitis B virus-DNA at separate timepoints. | 6, 12, 18, 24, 32, 48 and 60 month
  Measurement of decrease of hepatitis B virus-DNA and quota of patients with non-detectable hepatitis B virus-DNA at several timepoints after treatment with entecavir(Baraclude®) within 12 month.
Quota of patients with normalization of Alanine transaminase(ALT)-measurement in blood at separate timepoints | 6,12, 18, 24, 32, 48 and 60 month
  Quota of patients with normalization of Alanine transaminase(ALT)-measurement in blood will be checked at separate timepoints after treatment with entecavir(Baraclude®) within 12 month.
Quota of patients with hepatitis B viral protein loss, antibodies to the the hepatitis B 'e' antigen seroconversion, surface antigen of the Hepatitis-B-Virus loss and antibodies to the hepatitis B core antigen seroconversion at separate timepoints | 6,12, 18, 24, 32, 48 and 60 month
  Quota of patients with core antigen hepatitis B viral protein (HBeAg) loss, antibodies to the the hepatitis B 'e' antigen(anti-HBe) seroconversion, surface antigen of the Hepatitis-B-Virus(HBsAg) loss and antibodies to the hepatitis B core antigen(anti-HBs) seroconversion will be checked at separate timepoints after treatment with entecavir(Baraclude®) within 12 month.
Incidence of side effects | 60 month
  Incidence of appearance of side effects of after 12 month treatment with entecavir(Baraclude®)within whole study period of 60 month.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Trautwein, Professor MD, Principal Investigator — Department of Internal Medicine III, University Hospital Aachen
Locations (1):
- Department of Internal Medicin III, University Hospital Aachen, Aachen, North Rhine-Westphalia, Germany